CLINICAL TRIAL: NCT02540005
Title: Coagulation Disorders After Aneurysmatic Subarachnoid Haemorrhage
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Annukka Vahtera, MD, Tampere University Hospital
Other Study IDs: 230215-1
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Aneurysmatic Subarachnoid Haemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Aneurysmatic subarachnoid haemorrhage: Acute subarachnoid haemorrhage (confirmed by computed tomography, CT, or cerebrospinal fluid erythrocyte count over 1000 x 106/l) AND confirmed origin either with computed angiography (CTA) or digital subtraction angiography (DSA)
  Interventions: Other: ROTEM analysis
- Control patients: Elective craniotomy due to non-ruptured intracranial aneurysm
  Interventions: Other: ROTEM analysis

INTERVENTIONS:
Other: ROTEM analysis

SUMMARY:
The main purpose of this study is to analyse the on-going coagulation process after aSAH. For investigation the investigators use the rotational thromboelastometry (ROTEM) which is a point-of-care test using a variety of activators to provide a targeted and a dynamic analysis of coagulation cascade. This is a prospective, observational clinical study done in 16 aSAH patients treated in Tampere University Hospital intensive care unit and 16 control patients (elective craniotomy due to non-ruptured intracranial aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Acute subarachnoid haemorrhage (confirmed by computed tomography, CT, or cerebrospinal fluid erythrocyte count over 1000 x 106/l) AND confirmed origin either with computed angiography (CTA) or digital subtraction angiography (DSA)
* Onset of symptoms ≤ 12 hours
* Expected to stay 72 hours in the ICU

Exclusion Criteria:

* Pregnancy
* Any long-term anticoagulant medication, except for low-dose aspirin (<150 mg/day)
* Known active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute aneurysmal subarachnoid haemorrhage patients
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
ROTEM analysis: MCF (mm) by EXTEM activators | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland